CLINICAL TRIAL: NCT00002051
Title: Double Blind Study of Thymopentin Effects on Patients With HIV-1 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Immunobiology Research Institute (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 015E; H87-101
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-11

CONDITIONS: HIV Infections
Keywords: Thymopentin; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Thymopentin

INTERVENTIONS:
Drug: Thymopentin

SUMMARY:
Examine the ability of thymopentin (Timunox) to:

Reduce the amount and/or frequency of virus isolation. Stimulate the immune system and alter the clinical findings in patients infected with HIV who do not yet have AIDS.

ELIGIBILITY:
Inclusion Criteria

Concurrent Treatment:

Allowed:

* Aerosolized pentamidine.

Prior Medication:

Allowed:

* Aerosolized pentamidine.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* AIDS as defined by the CDC (except for those with HIV "wasting syndrome").
* Significant hepatic disease.
* Thrombocytopenia (< 75000 platelets/mm3).
* Abnormal chest x-ray (indicative of active disease (opportunistic infection)) within 30 days prior to entry.
* Hemophilia A or B or other hematologic disorders requiring current or previous administration of blood products.
* Known hypersensitivity to thymopentin.

Prior Medication:

Excluded within 30 days of study entry:

* Immunomodulatory or experimental therapy.
* Excluded within 90 days of study entry:
* Zidovudine (AZT).

Patients must not have:

* AIDS as defined by the CDC (except for those with HIV "wasting syndrome").
* Significant hepatic disease.
* Thrombocytopenia (< 75000 platelets/mm3).

Patients with the following conditions are included:

* Seropositive for HIV-1 (ELISA assay) confirmed by Western blot.
* HIV-1 p24 antigen must be detected in supernatant fluids from co-cultures of patient's peripheral blood monocytes (PBMC) on two separate occasions.
* HIV "wasting syndrome".
* Must voluntarily sign consent.

History of intravenous drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Immunobiology Research Institute, Annandale, New Jersey, United States